CLINICAL TRIAL: NCT03757897
Title: The Influence of Dexmedetomidine Hypnosis on Cerebrospinal Fluid (CSF) Volume, Brain Diffusion and 'Stiffness' Characteristics
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The investigators were unable to implement a MRI compatible EEG for use in human subjects (equipment and technical issues).
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000024166
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Cerebrospinal Fluid Pressure Increased
Keywords: dexmedetomidine
MeSH Terms: conditions — Intracranial Hypertension | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a preliminary interventional trial in which participants will serve as their own controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dexmedetomidine induced sleep patients (Experimental): All subjects will be measured for CSF volume, diffusion parameters and mechanical 'stiffness' of the brain during wakefulness and during sleep-induced with dexmedetomidine (DEXM).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The standard dosing of 1mcg/kg will be implemented over 10 minutes followed by a maintenance infusion of 0.2-1.0 titrated to a the target BIS (60-70) during the 20 minutes prior to MRI.
  Other Names: DEXM

SUMMARY:
The primary goal is to quantify cerebrospinal fluid (CSF) volume, diffusion characteristics and mechanical properties of brain tissue at two states of arousal.

DETAILED DESCRIPTION:
The primary goal is to quantify cerebrospinal fluid (CSF) volume, diffusion characteristics and mechanical properties of brain tissue at two states of arousal:

1. Resting, awake state
2. During sleep with low-dose intravenous infusion of dexmedetomidine (titrated to a Bispectral index (BIS) of 60-70)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Males or females between 18 and 40 years of age. Determined to be American Society of Anesthesiologist (ASA) 1 subjects.
2. Ability to provide written informed consent.

Exclusion Criteria:

1. Subjects with potential difficult airway as determined by the anesthesiologist
2. History of or family history of difficulty with anesthesia or sedation procedures
3. Known intolerance to dexmedetomidine
4. Body mass index >30
5. Subjects with any of the following: narcolepsy, obstructive sleep apnea (OSA) and/or abnormal sleeping patterns (including but not limited to those who use a Continuous positive Airway Pressure (C-PAP) machine, sleeping during the day, using medication to fall asleep, subjects reporting snoring as determined by self- report using Snoring, Tiredness, Observed apnea, Blood pressure, Body mass index, Age, Neck circumference and Gender (STOP-BANG) questionnaire (i) for undiagnosed OSA (3 or more 'yes' answers will exclude) and/or medical history;
6. Subjects with a history of restless leg syndrome as determined by self-report and/or medical history;
7. Use, in the past two weeks, of psychoactive medications (four weeks for fluoxetine) or medications that may affect brain function (including but not limited to opioid analgesics, antidepressants, antipsychotics, benzodiazepines and barbiturates) as determined by self-report and/or medical history;
8. Current or past Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnosis of a psychiatric disorder if it was severe enough to require the use of medications and or hospitalization to treat the condition.
9. Major medical problems that can impact brain function (e.g., problems of the Central Nervous System including seizures and psychosis; cardiovascular disease including hypertension and arrhythmias; metabolic, autoimmune, endocrine disorders) as determined by self-report, medical history and/or clinical exam;
10. Hepatic dysfunction or impairment as determined by subjects' self-reported history
11. Head trauma with loss of consciousness for more than 60 minutes as determined by self-report and/or medical history;
12. Positive urine test for controlled substances (cocaine, methamphetamine, amphetamines, opioids, cannabinoids, benzodiazepines and barbiturates) at the screening visit and at each visit of imaging study and neuropsychological assessment;
13. Positive urine pregnancy test;
14. Nursing mothers will be excluded
15. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (including but not limited to pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, large tattoos, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces as determined by the self-report checklist.
16. Fear of enclosed spaces (claustrophobia) as determined by self-report and medical history.
17. Cannot lie comfortably flat on the back for up to 3 hours in the MRI scanner as determined by self- report.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
CSF volume increase by 10% | 2 hours 30 minutes
  We hypothesize that CSF volume (as measured by T1 relaxation) will expand by 10% with DEXM- induced sleep compared to wakefulness. The increase in CSF volume during DEXM-induced sleep occurs because DEXM lowers central norepinephrine tone and sleep causes an increase in the interstitial fluid (ISF) volume (cell volume shrinks). MRI will take place 30 minutes after dexmedetomidine infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Benveniste, MD, PhD, Principal Investigator — Yale University